CLINICAL TRIAL: NCT06612853
Title: Cross-cultural Adaptation Into German and Italian, Validation, Reproducibility, and Responsiveness of the Single-item Sleep Quality Scale in Spine Patients
Brief Title: Validation of the Single-item Sleep Quality Scale
Acronym: SQS
Status: Recruiting | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: WS-0105
Record Dates: First submitted 2024-08-08; First posted 2024-09-25 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Spine Disorder
Keywords: Cross cultural adaptation; Translation; Validity; Reproducebility; Responsiveness; SQS; Sleep quality
MeSH Terms: conditions — Spinal Diseases; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pilot testing: A sample of n=20 Italian-speaking spine patients will complete the pre-final Italian version of the SQS and then be interviewed to discuss linguistic clarity and relevance. The same process will be performed with native German speakers for the German versions of the SQS
  Interventions: Other: Sleep Quality Scale (SQS)
- Field testing: A sample of n=100 Italian-speaking spine patients will complete the final translated Italian version of the SQS, together with the PSQI. The same process will be performed for n=100 German-speaking patients.
  Interventions: Other: Sleep Quality Scale (SQS); Other: Pittsburgh Sleep Quality Index (PSQI)

INTERVENTIONS:
Other: Sleep Quality Scale (SQS) — For the pilot testing, each patient will complete the pre-final version of the SQS.
  The patients involved in the field study will have to fill in the SQS twice before treatment, one week apart, to assess reproducibility of the scale and a third time at 3 months after treatment (surgical or conservative) to assess the responsiveness of the scale.
Other: Pittsburgh Sleep Quality Index (PSQI) — The patients involved in the field test will have to fill in the PSQI twice before treatment, one week apart, to assess reproducibility of the scale and a third time at 3 months after treatment (surgical or conservative) to assess the responsiveness of the scale.
  Groups: Field testing

SUMMARY:
The single-item sleep quality scale (SQS) allows patients to provide a self-assessment of sleep quality over a 7-day recall period without significant additional burden. However, the SQS has not yet been utilized or validated in patients with spine pathologies. The main purpose of this study is to cross-culturally adapt the SQS from English to German and Italian and to test its validity in patients with back disorders. The study will be conducted in two stages. The first stage will involve the translation and cross-cultural adaptation of the SQS from English to German and Italian. The second stage will involve the evaluation of the instrument's face, content, and construct validity, reproducibility, and responsiveness in patients with back disorders.

DETAILED DESCRIPTION:
Low back pain (LBP) consistently ranks as the leading cause of disability globally, prompting individuals affected by LBP to frequently seek healthcare. Utilizing reliable Patient-Reported Outcome Measures (PROMs) aids healthcare providers in assessing pain, functional impairment, disability, satisfaction, and quality of life in a standardized manner. However, the use of a validated questionnaire to assess each of these domains is not practicable in clinical practice. To solve this problem, the multidimensional Core Outcome Measures Index (COMI) was developed to assess the impact of LBP, using a brief set of questions. COMI has been demonstrated as a valuable metric when compared to alternative methods, exhibiting no significant limitations in terms of floor or ceiling effects and demonstrating outstanding construct validity. Moreover, it has also been established as a sensitive tool for assessing the perceived changes in patients following treatment. Recently, a complementary set of single-item measures to assess four of the "core" yellow flags (depression, anxiety, catastrophizing, and fear-avoidance) has been developed and defined as the "Core Yellow Flags Index" (CYFI). THE CYFI has been proven to be a valid and brief instrument for the assessment of key psychological factors in patients undergoing spine surgery and it also made a relevant contribution in predicting postoperative outcomes in this population. The brevity of the CYFI makes it a useful addition to the COMI in the self-assessment of baseline status before surgery.

Curiously, sleep has rarely been studied in this population and both the COMI and the CYFI do not evaluate this important variable. Assessing sleep in patients affected by spine disorders, including LBP, is of paramount importance due to the significant impact sleep disturbances can have on both the progression and management of these conditions. Sleep plays a crucial role in various physiological processes, including pain modulation, tissue repair, immune function, and psychological well-being. Therefore, disruptions in sleep patterns can exacerbate symptoms, impair recovery, and diminish the overall quality of life for individuals with back disorders. Recognizing the substantial impact of sleep-related challenges on individuals and their consequential implications, it becomes crucial to employ tools for assessing sleep quality in clinical settings.

Sleep assessment involves the measurement of various parameters, including sleep duration, sleep architecture, sleep latency, and the frequency and duration of nocturnal awakenings. Objective methods such as polysomnography (PSG) and/or actigraphy, or the use of sleep-rating questionnaires, are typically employed to quantitatively assess these metrics. The established benchmark for evaluating sleep quality continues to be PSG and/or electroencephalographic spectral analysis, despite the effectiveness of behavioural parameters in certain contexts, such as actigraphy. However, both PSG and EEG analyses may pose logistical challenges in large-scale and field studies. To address these constraints and to obtain preliminary insights into potential sleep disorders in different populations, several sleep questionnaires have been formulated and validated. Despite their efficacy in gauging sleep quality, these tools exhibit limitations when applied in clinical trials. A case in point is the Pittsburgh Sleep Quality Index (PSQI), a commonly utilized measure for assessing sleep quality, since its extended format incorporating 19 rating items may render it impractical for administration to participants in clinical trials. Further, the PSQI exhibits limitations due to its utilization of only four potential response levels for the sleep quality question. This constraint could restrict respondents when assigning grades to their sleep quality, potentially compromising the precision of their responses. Moreover, such a limited scale may fail to capture minor or nuanced changes in sleep quality. Consequently, despite the existence of alternative sleep quality questionnaires, there persists a requirement to create and validate innovative instruments explicitly tailored for assessing sleep quality in the framework of clinical trials. These novel questionnaires should address the shortcomings associated with response level constraints to enhance the accuracy and sensitivity of sleep quality evaluations in research settings.

Recently, the single-item sleep quality scale (SQS) was developed as a simple and practical sleep quality assessment. The authors reported that the SQS possesses excellent concurrent criterion validity and strong correlations between the SQS and the sleep quality items of the PSQI in patients with insomnia were detected. The SQS represents a pragmatic advancement in sleep quality assessment within clinical settings, distinguishing itself from conventional standards. Developed as a self-rated global tool, SQS offers an efficient approach based on a comprehensive review of pertinent sleep quality aspects, incorporating critical components from the PSQI, and incorporating expert and patient feedback. The single-item format permits patients to provide a self-assessment of sleep quality over a 7-day recall period without significant additional burden. Employing a visual analogue scale (VAS) enhances the potential for a more sensitive measurement, contributing to the utility of SQS in capturing nuanced variations in sleep quality. This innovation addresses the need for a streamlined yet effective tool for sleep quality evaluation in clinical contexts. However, the SQS has not yet been adapted for the German and Italian languages, nor it has been validated in spine patients.

Regarding risk category, the project shall be identified as Category A (only minimal risk and burden regarding the planned measures for sampling biological material or collecting personal data). The rationale for the categorization is based on the study objectives and study design.

This project will be carried out in accordance with the protocol and with principles enunciated in the current version of the Declaration of Helsinki, the guidelines of Good Clinical Practice (GCP) issued by ICH, in case of medical device: the European Directive on medical devices 93/42/EEC and the ISO Norm 14155 and ISO 14971, the Swiss Law and Swiss regulatory authority's requirements. The approval will be sought from the local responsible independent Competent Ethics Committee (CEC) in Zurich. In accordance with GCP, the project will be implemented only after obtaining approval for this protocol, and other study-specific documents by the local responsible independent CEC. Participants consenting to participate in the study will be enrolled. The CEC will be informed about study stop/end in agreement with local requirements.

ELIGIBILITY:
Inclusion Criteria:

* both male and female patients
* German-speaking or Italian-speaking
* diagnosis of spine pathology
* age ≥ 14 years
* cognitively intact (self-reported)

Exclusion Criteria:

* pregnancy (self-reported)
* medical and/or pharmacological treatment for sleep disorders
* melatonin intake
* daily use of smart-watch or applications for automatic sleep detection
* inability to give informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with spinal disorders, being considered for spinal surgery or conservative treatment, and with a good understanding of the German or Italian language will be recruited at the Schulthess Clinic. For the pilot testing, patients will be recruited immediately after their outpatient examination. For the field testing, patients waiting for surgery or conservative treatment will be recruited. A total of 20 patients, complying with the inclusion and exclusion criteria listed above, will be involved in the pilot test and a total of 100 patients will be involved in the field test. Therefore, n=120 patients will be recruited for each language translation, with a total of n=240 patients.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Translation and cross-cultural adaptation of the Single-item Sleep Quality Scale (SQS) in Italian and German | Within 8 weeks following the enrollment of the translators and expert commitee for the translation process.
  Outcome: translated version of the SQS in Italian and German
Field-testing of the Single-item Sleep Quality Scale (SQS) final translated version for responsiveness | At 3 months (week 12) after treatment (surgical or conservative)
  SQS responsiveness. A ROC curve analysis will be used to explore the ability of the SQS change scores to differentiate between patients who have and have not improved (dichotomized), according to the Pittsburgh Sleep Quality Index (PSQI) delta scores of Item 6 (sleep quality). Using the ROC curve, the responsiveness will be described in terms of sensitivity and specificity. We will consider an AUC of at least 0.70 to be adequate. The optimal cut off point will be computed using the Youden index.
Field-testing of the Single-item Sleep Quality Scale (SQS) final translated version for construct validity | At week 1, before treatment.
  SQS construct validity. Outcome: the construct validity will be calculated through Spearman's correlation coefficient between SQS score (from 0 to 10) and the questionnaire item 6 (sleep quality) of the Pittsburgh Sleep Quality Index (PSQI).
  The strength of the relationship will be described as excellent (0.81-1.0), very good (0.61-0.80), good (0.41-0.60), fair (0.21-0.40), and poor (0.20-0.0).
Pilot-testing of the Single-item Sleep Quality Scale (SQS) pre-final translated version for content validity | Within 8 weeks from the enrollment of the patients. Patients will be recruited immediately after their outpatient examination and they will fill in the SQS once.
  SQS content validity Outcome: the content validity ratio (CVR). CVR will be calculated as follows: CVR= [ne - (N/2)] / (N/2), where ne is the number of experts indicating an item "essential," and N is the total number of experts. Therefore, considering the sample size (n=20) for pilot testing and the recognized Lawshe's CVR critical values, a CVR value of 0.50 is expected (corresponding to a 75% of agreement).

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mannion AF, Porchet F, Kleinstuck FS, Lattig F, Jeszenszky D, Bartanusz V, Dvorak J, Grob D. The quality of spine surgery from the patient's perspective. Part 1: the Core Outcome Measures Index in clinical practice. Eur Spine J. 2009 Aug;18 Suppl 3(Suppl 3):367-73. doi: 10.1007/s00586-009-0942-8. Epub 2009 Mar 25. PMID 19319578
- [Background] Mannion AF, Mariaux F, Reitmeir R, Fekete TF, Haschtmann D, Loibl M, Jeszenszky D, Kleinstuck FS, Porchet F, Elfering A. Development of the "Core Yellow Flags Index" (CYFI) as a brief instrument for the assessment of key psychological factors in patients undergoing spine surgery. Eur Spine J. 2020 Aug;29(8):1935-1952. doi: 10.1007/s00586-020-06462-z. Epub 2020 Jun 16. PMID 32556625
- [Background] Szentkiralyi A, Madarasz CZ, Novak M. Sleep disorders: impact on daytime functioning and quality of life. Expert Rev Pharmacoecon Outcomes Res. 2009 Feb;9(1):49-64. doi: 10.1586/14737167.9.1.49. PMID 19371179
- [Background] Littner M, Kushida CA, Anderson WM, Bailey D, Berry RB, Davila DG, Hirshkowitz M, Kapen S, Kramer M, Loube D, Wise M, Johnson SF; Standards of Practice Committee of the American Academy of Sleep Medicine. Practice parameters for the role of actigraphy in the study of sleep and circadian rhythms: an update for 2002. Sleep. 2003 May 1;26(3):337-41. doi: 10.1093/sleep/26.3.337. PMID 12749556
- [Background] Littner M, Hirshkowitz M, Kramer M, Kapen S, Anderson WM, Bailey D, Berry RB, Davila D, Johnson S, Kushida C, Loube DI, Wise M, Woodson BT; American Academy of Sleep Medicine; Standards of Practice Committe. Practice parameters for using polysomnography to evaluate insomnia: an update. Sleep. 2003 Sep;26(6):754-60. doi: 10.1093/sleep/26.6.754. PMID 14572131
- [Background] Krystal AD, Edinger JD. Measuring sleep quality. Sleep Med. 2008 Sep;9 Suppl 1:S10-7. doi: 10.1016/S1389-9457(08)70011-X. PMID 18929313
- [Background] Lomeli HA, Perez-Olmos I, Talero-Gutierrez C, Moreno CB, Gonzalez-Reyes R, Palacios L, de la Pena F, Munoz-Delgado J. Sleep evaluation scales and questionaries: a review. Actas Esp Psiquiatr. 2008 Jan-Feb;36(1):50-9. PMID 18286400
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Snyder E, Cai B, DeMuro C, Morrison MF, Ball W. A New Single-Item Sleep Quality Scale: Results of Psychometric Evaluation in Patients With Chronic Primary Insomnia and Depression. J Clin Sleep Med. 2018 Nov 15;14(11):1849-1857. doi: 10.5664/jcsm.7478. PMID 30373688